CLINICAL TRIAL: NCT01340326
Title: The Impact of Dose of Angiotensin-receptor Blocker Valsartan and Genetic Polymorphism on the Post-MI Ventricular Remodeling
Acronym: VALID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Kyungil Park, Assistant professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Donga 419
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Myocardial Infarction
Keywords: Post myocardial infarction ventricular remodeling; valsartan
MeSH Terms: conditions — Myocardial Infarction | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valsartan,high dose (Active Comparator): high dose group (valsartan up to 320 mg/day)
  Interventions: Drug: high dose of valsartan
- Valsartan, usual dose (Other): usual dose group (valsartan 80 mg/day)
  Interventions: Drug: usual dose of valsartan

INTERVENTIONS:
Drug: high dose of valsartan — comparison of different dosages of drug
  Arms: Valsartan,high dose
Drug: usual dose of valsartan — comparison of different dosages of drug
  Arms: Valsartan, usual dose

SUMMARY:
Angiotensin-converting enzyme inhibitors and angiotensin-receptor blocker valsartan ameliorate ventricular remodeling after myocardial infarction (MI). Although the amount of those drugs used in previous clinical trials, therefore recommended in practical guidelines is maximum clinical dose, it has not been clearly demonstrated whether the recommended dose is more efficacious compared to lower dose commonly used in clinical practice. In addition, the impact of genetic polymorphism in neurohormonal system on the pharmacological effect has not been explored in the setting of post-MI remodeling.

Therefore, the investigators evaluate whether submaximal dose, which are lower than those in major pivotal trials but typically used in clinical practice, can offer similar benefit in post-MI ventricular remodeling.

DETAILED DESCRIPTION:
A total of 1116 patients with left ventricular (LV) dysfunction following the first episode of acute ST-elevation MI are to be enrolled and randomized to maximal tolerable dose (up to 320 mg/day) or usual dose (80 mg/day) of valsartan for 12 months in 2:1 ratio. Echocardiographic analysis for quantifying post-MI ventricular remodeling and genotyping of blood samples are conducted in central core laboratory. Clinical assessment and laboratory test are performed at fixed times, and genetic polymorphisms of the patients are tested at the time of admission.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age > 18
* First episode of acute ST-elevation MI
* An echocardiographic left ventricular ejection fraction less than 50 %
* Patients who provide written informed consent

Exclusion Criteria:

* Contraindications for use of angiotensin receptor blockers (ARBs)(hypersensitivity, pregnancy, bilateral renal artery stenosis)
* Urgent need for revascularization procedure
* Severe heart failure (need for intravenous inotropic support)
* Persistent (> 1 hour) severe hypotension (systolic blood pressure < 90 mmHg)
* Refractory or potentially lethal arrhythmias
* Hemodynamically significant right ventricular infarction
* Primary valvular diseases
* Congenital heart disease
* Idiopathic hypertrophic cardiomyopathy
* Concomitant inflammatory cardiopathy
* Significant hepatic dysfunction
* Significant renal dysfunction
* Anemia (hemoglobin < 10 mg/mL)
* Psychiatric disorders, alcohol or durg abuse
* Any concomitant disease that might interfere with drug evaluation (especially if life expectancy is less than 1 year)
* Participation in any other pharmacological study within 2 months
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2007-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the left ventricular volume index from baseline to follow-up | at 24hrs, 1month, and 12months after myocardial infarction
  We measured a left ventriular volume index by echocardiography.
left ventricular volume index | at 12months after myocardial infarction

SECONDARY OUTCOMES:
clinical events | during 12 months follow up
  Clinical events were defined as all cause death and hospitalization due to cardiovascular problems.
clinical events | at 12 months after myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine,Dong-A University College of Medicine, Busan, South Korea

REFERENCES:
- [Derived] Cho YR, Kim YD, Park TH, Park K, Park JS, Baek H, Choi SY, Kim KS, Hong TJ, Yang TH, Hwang JY, Park JS, Hur SH, Lee SG. The impact of dose of the angiotensin-receptor blocker valsartan on the post-myocardial infarction ventricular remodeling: study protocol for a randomized controlled trial. Trials. 2011 Nov 22;12:247. doi: 10.1186/1745-6215-12-247. PMID 22108275